CLINICAL TRIAL: NCT00036868
Title: A Randomized Phase II Study Of CMF Alone And In Combination With Anti c-erbB2 Antibody (Herceptin) In Women With c-erbB2 Positive Metastatic Breast Cancer
Brief Title: Combination Chemotherapy With Trastuzumab in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-10995-16999; EORTC-10995; EORTC-16999; IDBBC-EORTC-10995
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; CMF regimen; Cyclophosphamide; Fluorouracil; Methotrexate

ARMS (1):
- CMF + Herceptin (Experimental)
  Interventions: Biological: trastuzumab; Drug: CMF regimen; Drug: cyclophosphamide; Drug: fluorouracil; Drug: methotrexate

INTERVENTIONS:
Biological: trastuzumab
Drug: CMF regimen
Drug: cyclophosphamide
Drug: fluorouracil
Drug: methotrexate

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as cyclophosphamide, methotrexate, and fluorouracil use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy with trastuzumab may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining combination chemotherapy with trastuzumab in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence of clinical heart failure in women with c-erbB2-positive metastatic breast cancer treated with cyclophosphamide, methotrexate, and fluorouracil in combination with trastuzumab (Herceptin®).
* Compare the therapeutic activity of this regimen, in terms of objective response rate, in these patients.
* Compare the duration of response and time to progression in patients treated with this regimen.
* Compare the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive CMF comprising cyclophosphamide orally on days 1-14 or IV on days 1 and 8 and methotrexate IV and fluorouracil IV on days 1 and 8. Patients also receive trastuzumab (Herceptin®) IV over 30-90 minutes once weekly beginning on day 1. Treatment repeats every 4 weeks for 8 courses. Patients then receive trastuzumab once every 3 weeks in the absence of disease progression, unacceptable toxicity, or patient refusal.

Patients are followed every 8 weeks until documentation of disease progression or initiation of a new anticancer therapy. Patients developing disease progression are followed every 12 weeks.

PROJECTED ACCRUAL: A total of 66 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast cancer c-erbB2 positive (3+ overexpression by the HercepTest™ method) in the primary tumor or metastatic site
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * Lesions that have been irradiated in the preceding 3 months cannot be used as target lesions unless they have appeared or clearly progressed since prior irradiation
  * No bone lesions as the only target lesions
* No contralateral breast cancer that is c-erbB2-positive or c-erbB2-negative/unknown, with status determined on a metastatic site
* No CNS metastases

  * CT scan of brain and CSF cytology are required if neurologic symptoms are present
* Hormone receptor status:

  * Any estrogen or progesterone receptor status

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Any status

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* Transaminases less than 2.5 times ULN (5 times ULN if liver metastases present)

Renal:

* For patients age 18 to 69:

  * Creatinine no greater than ULN
* For patients age 70 and over:

  * Creatinine clearance normal

Cardiovascular:

* LVEF normal by MUGA or echocardiogram
* No clinical heart failure

Pulmonary:

* No malignancy-associated dyspnea at rest
* No requirement for supportive oxygen therapy

Other:

* Not pregnant or nursing
* No other prior or concurrent malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude compliance with study therapy and follow-up schedule

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior anti-c-erbB2 antibody, including trastuzumab (Herceptin®)
* No other concurrent biologic therapy

Chemotherapy:

* No more than 1 prior chemotherapy regimen for metastatic breast cancer
* Prior combination of cyclophosphamide, methotrexate, and fluorouracil (CMF) allowed in the adjuvant or metastatic setting only if the disease-free interval after completion of CMF was at least 12 months
* Prior anthracyclines and/or taxanes allowed
* At least 4 weeks since prior anthracyclines
* No prior cumulative dose of doxorubicin more than 360 mg/m^2
* No prior cumulative dose of epirubicin more than 720 mg/m^2
* No prior cumulative dose of mitoxantrone more than 90 mg/m^2
* No other concurrent chemotherapy

Endocrine therapy:

* More than 2 weeks since prior hormonal therapy in the adjuvant or metastatic setting
* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent anticancer therapy or investigational drugs
* No concurrent bisphosphonates started after study enrollment except for hypercalcemia

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-02; Primary Completion 2009-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Clinical heart failure rate measured by New York Heart Association classification, LVEF, and ECG | from registration
Response rate by RECIST | from registration

SECONDARY OUTCOMES:
Duration of response by RECIST | from registration
Time to progression | from registration
Toxicity measured by CTC v2.0 | from registration

CONTACTS AND LOCATIONS:
Overall Officials: David Cameron, Study Chair — Western General Hospital, Edinburgh
Locations (13):
- Belgium (3):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
- Herlev Hospital - University Hospital of Copenhagen, Copenhagen, Denmark
- National Cancer Institute of Egypt, Cairo, Egypt
- Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon, France
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen
- Medical University of Gdansk, Gdansk, Poland
- Institute of Oncology and Radiology of Serbia, Belgrade, Serbia
- Medical Oncology Centre of Rosebank, Johannesburg, South Africa
- Western Infirmary, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] Neskovic-Konstantinovic Z, Nooij M, Khaled H, et al.: Safety and efficacy of combined trastuzumab and CMF therapy in women with metastatic breast cancer: EORTC protocol 10995. [Abstract] J Clin Oncol 25 (Suppl 18): A-1040, 2007.
- [Derived] Tryfonidis K, Marreaud S, Khaled H, De Valk B, Vermorken J, Welnicka-Jaskiewicz M, Aalders K, Bartlett JMS, Biganzoli L, Bogaerts J, Cameron D; EORTC- Breast Cancer Group. Cardiac safety, efficacy, and correlation of serial serum HER2-extracellular domain shed antigen measurement with the outcome of the combined trastuzumab plus CMF in women with HER2-positive metastatic breast cancer: results from the EORTC 10995 phase II study. Breast Cancer Res Treat. 2017 Jun;163(3):507-515. doi: 10.1007/s10549-017-4203-y. Epub 2017 Mar 21. PMID 28324265